CLINICAL TRIAL: NCT02579967
Title: Pilot Trial of Allogeneic Blood or Marrow Transplantation for Primary Immunodeficiencies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160003; 16-C-0003
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01-16

CONDITIONS: Primary T-cell Immunodeficiency Disorders; Common Variable Immunodeficiency; Immune System Diseases; Autoimmune Lymphoproliferative; Lymphoproliferative Disorders
Keywords: Haploidentical; Autoimmunity; Immune Dysregulation; Congenital; Opportunistic Infection
MeSH Terms: conditions — T cell immunodeficiency primary; Common Variable Immunodeficiency; Immune System Diseases; Lymphoproliferative Disorders; Autoimmune Diseases; Opportunistic Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1/ IOC Arm-Closed with amendment L (07/05/2019) (Experimental): Immunosuppression Only Conditioning Arm
  Interventions: Drug: Immunosuppression Only Conditioning -Closed with amendment L; Drug: GVHD Prophylaxis; Procedure: Allo BMT
- 2/ RIC Arm - Closed with Amendment L (07/05/2019) (Experimental): Reduced Intensity Conditioning Arm
  Interventions: Drug: Reduced Intensity Conditioning; Drug: GVHD Prophylaxis; Procedure: Allo BMT
- 3/ MAC Arm-Closed with amendment L (07/05/2019) (Experimental): Myeloablative Conditioning Arm
  Interventions: Drug: Myeloablative Conditioning-Closed with amendment L; Drug: GVHD Prophylaxis; Procedure: Allo BMT
- 4/ RIC-MMF Arm (Experimental): Reduced Intensity Conditioning with MMF duration de-escalation design
  Interventions: Drug: Reduced Intensity Conditioning; Drug: GVHD Prophylaxis; Procedure: Allo BMT
- 5/ Donor Arm (No Intervention): Donor
- 6/ RIC-SHORT Arm (Experimental): Reduced Intensity Conditioning with shortened duration and dose-reduced PTCy
  Interventions: Drug: Reduced Intensity Conditioning; Drug: GVHD Prophylaxis; Procedure: Allo BMT

INTERVENTIONS:
Drug: Immunosuppression Only Conditioning -Closed with amendment L — Pentostatin 4 mg/m2/day IV on days -9 and -5, cyclophosphamide 5 mg/kg orally daily on days -9 through -2 (Closed with amendment L)
  Arms: 1/ IOC Arm-Closed with amendment L (07/05/2019)
Drug: Reduced Intensity Conditioning — pentostatin 4 mg/m2/day IV on days -11 and -7, cyclophosphamide 3 mg/kg orally daily on days -11 through -4; busulfan IV, pharmokinetically dosed, on days -3 and -2.
  Arms: 2/ RIC Arm - Closed with Amendment L (07/05/2019); 4/ RIC-MMF Arm; 6/ RIC-SHORT Arm
Drug: Myeloablative Conditioning-Closed with amendment L — Pentostatin 4 mg/m2/day IV on days -13 and -9, low-dose cyclophosphamide orally daily on days -13 through -6; busulfan IV, pharmokinetically dosed, on days -5, -4, -3, and -2. (Closed with amendment L)
  Arms: 3/ MAC Arm-Closed with amendment L (07/05/2019)
Drug: GVHD Prophylaxis — High-dose, post-transplantation cyclophosphamide (PTCy) 25-50 mg/kg on days +3 and +4, sirolimus 6 mg on days +5 through +90, and mycophenolate mofetil (MMF) on days +5 through 0, +18, +25, or +35 depending on treatment arm and cohort.
  Arms: 1/ IOC Arm-Closed with amendment L (07/05/2019); 2/ RIC Arm - Closed with Amendment L (07/05/2019); 3/ MAC Arm-Closed with amendment L (07/05/2019); 4/ RIC-MMF Arm; 6/ RIC-SHORT Arm
Procedure: Allo BMT — Allogeneic blood or marrow transplantation
  Arms: 1/ IOC Arm-Closed with amendment L (07/05/2019); 2/ RIC Arm - Closed with Amendment L (07/05/2019); 3/ MAC Arm-Closed with amendment L (07/05/2019); 4/ RIC-MMF Arm; 6/ RIC-SHORT Arm

SUMMARY:
Background:

Allogeneic blood or marrow transplant is when stem cells are taken from one person s blood or bone marrow and given to another person. Researchers think this may help people with immune system problems.

Objective:

To see if allogeneic blood or bone marrow transplant is safe and effective in treating people with primary immunodeficiencies.

Eligibility:

Donors: Healthy people ages 4 or older

Recipients: People ages 4-75 with a primary immunodeficiency that may be treated with allogeneic blood or marrow transplant

Design:

Participants will be screened with medical history, physical exam, and blood tests.

Participants will have urine tests, EKG, and chest x-ray.

Donors will have:

Bone marrow harvest: With anesthesia, marrow is taken by a needle in the hipbone.

OR

Blood collection: They will have several drug injections over 5-7 days. Blood is taken by IV in one arm, circulates through a machine to remove stem cells, and returned by IV in the other arm.

Possible vein assessment or pre-anesthesia evaluation

Recipients will have:

Lung test, heart tests, radiology scans, CT scans, and dental exam

Possible tissue biopsies or lumbar puncture

Bone marrow and a small piece of bone removed by needle in the hipbone.

Chemotherapy 1-2 weeks before transplant day

Donor stem cell donation through a catheter put into a vein in the chest or neck

Several-week hospital stay. They will take medications and may need blood transfusions and additional procedures.

After discharge, recipients will:

Remain near the clinic for about 3 months. They will have weekly visits and may require hospital readmission.

Have multiple follow-up visits to the clinic in the first 6 months, and less frequently for at least 5 years.

DETAILED DESCRIPTION:
Background:

* Primary immunodeficiency diseases (PIDs) are conditions associated with major quantitative or qualitative immunologic abnormalities that are, in most cases, due to defects in cells of hematopoietic origin
* Participants with PID can have life-threatening complications including malignancy, recurrent infection, and autoimmunity/immune dysregulation
* Allogeneic blood or marrow transplantation (allo BMT) has the potential to cure the immune defect in PID and thereby reduce the morbidity and mortality associated with these diseases

Objectives:

-To estimate the acute graft-versus-host disease (aGVHD)-free, graft failure-free survival at day +180 after allo BMT, analyzed separately by conditioning arm/cohort

Eligibility:

* Patients age >= 4 through 75 years
* PID deemed to be of sufficient past severity to warrant allo BMT, by meeting the two criteria below:

  * PID as defined by identified genetic defect or, in the absence of a mutation, patients with an immune defect potentially amenable to allo BMT who meet the clinical history criteria below may be eligible
  * Clinical history of at least two of the following:

    * Life-threatening, organ-threatening, or severely disfiguring infection
    * Protracted or recurrent infections
    * Infection with an opportunistic organism
    * Chronic elevation in the blood of a latent virus
    * Evidence of immune dysregulation
    * Hypogammaglobulinemia/dysglobulinemia
    * Hematologic malignancy or lymphoproliferative disorder
    * Virus-associated solid tumor malignancy or pre-cancerous lesion
* At least one 7-8/8 (9-10/10) HLA-matched related or unrelated donor, or an HLA-haploidentical related donor
* Adequate end-organ function
* Consensus opinion by the investigative team that the patient has the potential to benefit from transplant despite existing, non-hematopoietic organ dysfunction
* Not pregnant or breastfeeding
* HIV negative
* Disease status: patients with malignancy should be referred in remission for evaluation, except in the case of virus-associated malignancy who may be referred at any time

Design:

* The study will have two arms that vary in mycophenolate mofetil (MMF) duration.
* RIC and RIC-MMF arms: pentostatin 4 mg/m2/day IV on days -11 and -7, low-dose cyclophosphamide orally daily on days -11 through -4; busulfan IV, pharmacokinetically dosed, on days -3 and -2.
* RIC-SHORT arm: pentostatin 4 mg/m2/day IV on days -9 and -5, low-dose cyclophosphamide orally daily on days -9 through -2; busulfan IV, pharmacokinetically dosed, on days -3 and -2.
* Bone marrow is the preferred graft source. Peripheral blood stem cells are permitted on RIC-MMF arm but not on RIC-SHORT arm.
* GVHD prophylaxis:

  * High-dose, post-transplantation cyclophosphamide (PTCy) on days +3 and +4, sirolimus on days +5 through +90, and mycophenolate mofetil (MMF) on days +5 through +35 for all arms except the RIC-MMF and RIC-SHORT arm. The RICMMF arm will receive MMF of varying durations based on a duration de-escalation schema.
  * RIC-SHORT: Reduced-dose, post-transplantation cyclophosphamide (PTCy) on days +3 and +4, sirolimus on days +5 through +90, and mycophenolate mofetil (MMF) on days +5 through +18 for all arms.

ELIGIBILITY:
* INCLUSION CRITERIA - RECIPIENT:
* Patients age >= 4 through 75 years
* PID deemed to be of sufficient past severity to warrant allo BMT, by meeting the two criteria below:

  1. PID as defined by identified genetic defect or, in the absence of a PID-associated genetic mutation, patients with an immune defect potentially amenable to allo BMT who meet the clinical history criteria below may be eligible upon discussion with the PI

     * Mutations should be confirmed in a CLIA-certified laboratory, if such testing is available.
     * Patients without a mutation must be deemed eligible and appropriate for allo BMT by the PI. Some patients may meet the clinical history criteria listed below, but will not be eligible if it is thought that their clinical history is due to a condition apart from an immune defect. In addition, patients with a PID of mild severity, such as those with selective IgA deficiency, may meet at least two of the clinical history criteria, but may be deemed inappropriate for allo BMT by the PI if it is felt that the risks of the procedure outweigh the severity of the disease.
  2. Clinical history of at least two of the following:

     * Life-threatening, organ-threatening, or severely disfiguring infection
     * Protracted or recurrent infections requiring unusually long or repeated courses of antibiotics
     * Infection with an opportunistic organism
     * Chronic elevation in the blood (>=2 documented elevations over a period of 6 months or longer) of a latent virus (EBV, CMV, HHV6, HHV8, etc.)
     * Evidence of immune dysregulation, as manifested by autoimmune disease, atopy, hemophagocytic lymphohistiocytosis/macrophage activation syndrome, granulomas, splenomegaly, or lymphadenopathy
     * Patients with hemophagocytic lymphohistiocytosis or macrophage activation syndrome related to an underlying lymphoma with no other clinical history suggestive of a primary immunodeficiency will not be eligible
     * Hypogammaglobulinemia, dysglobulinemia, or impaired response to vaccination
     * Hematologic malignancy or lymphoproliferative disorder
     * Tissue diagnosis should be confirmed by NCI Department of Pathology, if prior biopsies are available
     * Virus-associated solid tumor malignancy or pre-cancerous lesion
     * Tissue diagnosis should be confirmed by NCI Department of Pathology, if prior biopsies are available
* Availability of at least one 7-8/8 (9-10/10) HLA-matched related (excluding an identical twin) or unrelated donor, or an HLA-haploidentical related donor
* Consensus among the PI, key AIs, and consultants (as necessary) that correction of the patient s immune system through BMT has the potential to improve the patient s health, quality of life, and/or life expectancy, after taking into consideration the patient s existing non-hematopoietic, potentially irreversible organ dysfunction
* Adequate end-organ function, as measured by:

  * Left ventricular ejection fraction (LVEF) >= 40% by 2D echocardiogram (ECHO) or MUGA, or left ventricular shortening fraction >= 20% by ECHO for patients receiving RIC or RIC-MMF, or RIC-SHORT, or LVEF >= 30% if the patient has radiologic evidence of aortic, renal, or coronary artery vasculitis.
  * Pulmonary function tests: DL(co) (corrected for hemoglobin) and FEV(1) >= 40% of predicted for the RIC, RIC-MMF, and RIC-SHORT arms; or in pediatric patients, if unable to perform pulmonary function tests, there should be no evidence of dyspnea at rest, no requirement for supplemental oxygen, and oxygen saturation >92% on room air. Calculations will be based on the values reported in CRIS.
  * Bilirubin <= 3.0 mg/dL (unless due to Gilbert s syndrome or hemolysis) for patients receiving RIC, RIC-MMF, RIC-SHORT; ALT and AST 10 x ULN for patients receiving RIC, RIC-MMF, RIC-SHORT. Patients who are above these bilirubin, ALT, or AST thresholds may be eligible for the RIC, RIC-MMF, or RIC-SHORT arms if evaluated by a hepatologist who deems the liver function test abnormalities to be potentially reversible with bone marrow transplant.
  * Estimated creatinine clearance of >= 40 mL/min/1.73 m^2, calculated using the Cockcroft-Gault equation for adults and Schwartz formula for pediatric patients, for patients with creatinine levels above the institutional upper limit of normal
* Karnofsky or Lansky performance status of >=60% or ECOG performance status of 2 or less
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document
* Not pregnant or breastfeeding. As therapeutic agents used in this trial may be harmful to a fetus, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least one year post-allo BMT. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in the study, she should inform her treating physician immediately.
* Disease status: Patients with malignancy are to be referred in remission for evaluation, except in cases of virus-associated malignancy who may be referred at any time. Should a patient have progressive disease or a donor becomes unavailable after enrollment, the patient will be referred back to his/her primary hematologist-oncologist for treatment. If this course of action is not in the best interest of the patient according to the clinical judgment of the PI, then the patient may receive standard treatment for the malignant disease under the current study, although this should only occur as a bridge to transplant. If under either of these settings, it becomes apparent that the patient will not be able to proceed to transplant, then he/she must come off the study. Patients receiving standard therapy will be told about the therapy, associated risks, potential benefits, alternatives to the proposed therapy, and the availability of receiving the same treatment elsewhere, outside of a research protocol.

EXCLUSION CRITERIA - RECIPIENT:

* Patients who are receiving any other investigational agents, with the exception of virus-specific cytotoxic T-cells for the treatment of viral infection/reactivation prior to allo BMT.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents (cyclophosphamide, busulfan, pentostatin, sirolimus, MMF, filgrastim or filgrastim biosimilar) used in the study
* Active psychiatric disorder which may compromise compliance with the transplant protocol, or which does not allow for appropriate informed consent
* Active central nervous system (CNS) involvement by malignancy, except in cases of virus-associated malignancies with CNS involvement in which case the patient may benefit from the transplant to control the malignancy.
* MAGT1 mutation and active need to take anti-platelet agents and/or therapeutic anti-coagulation that cannot be interrupted during aplasia.
* HIV positive or other acquired immunodeficiency that, as determined by the PI, interferes with the assessment of PID severity and/or the attribution of clinical manifestations of immunodeficiency to a PID.
* Lack of adequate central venous access potential

Inclusion Criteria (Related Donor):

* Ages >= 4
* Related donor deemed suitable and eligible and willing to donate per clinical evalations who are additionally willing to donate blood, urine, and marrow specimens for research. Related donors will be evaluated in accordance with existing Standard Policies and Procedures for determination of eligibility and suitability for clinical donation. Note that participation in this study is offered to all related donors but is not required for clinical donation, so it is possible that not all related donors will enroll on this study.

Exclusion Criteria (Related Donor):

None

INCLUSION CRITERIA - UNRELATED DONOR:

* Ages >= 18
* Unrelated donors will be evaluated in accordance with existing NMDP Standard Policies and Procedures, available at: http://bethematch.org/About-Us/Global-transplant-network/Standards/, except for the additional requirement of EBV serostatus testing. Note that participation in this study is offered to all unrelated donors but not required for clinical donation, so it is possible that not all unrelated donors will enroll on this study.

EXCLUSION CRITERIA - UNRELATED DONOR:

-Unrelated donors: failure to qualify as a National Marrow Donor Program (NMDP) donor per current NMDP Standards, available at: http://bethematch.org/About-Us/Global-transplant-network/Standards/.

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2015-11-19 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
For the RIC-SHORT arm: To estimate the aGVHD-free, graft failure-free survival | +180 after allo BMT
  Proportion of participants without GVHD
For the RIC : To estimate the aGVHD-free, graft failure-free survival | +180 after allo BMT
  Proportion of participants without GVHD
For the RIC-MMF arm: To determine the shortest duration of MMF that can be safely administered without excessive rates of graft failure or acute grade 3-4 GVHD | Duration de-escalation design
  Shortest duration of MMF

SECONDARY OUTCOMES:
Transplant-related mortality | +180 and 1 year post transplant
  Cumulative incidence of transplant-related mortality at 180 days and 1 year post transplant.
Secondary graft failure | 1 year post transplant
  Cumulative incidence of secondary graft failure at 1 year post transplant.
Overall survival | 1 year post transplant
  Time from transplant to death of any cause.
Kinetics and durability of lineage-specific donor chimerism | days +28 and +42
  Median amount of patient who has early chimerism
Kinetics and durability of engraftment | days +28, +42, +60, +100, +180, and 1 year after allo BMT
  The percentage of donor T-, B-, NK-, and myeloid cell populations at days +28, +42, +60, +100, +180, and 1 year post transplant.
Incidence of Chronic Graft-versus-host disease | 1 and 2 years post transplant
  Cumulative incidence of chronic graft versus host disease at 1 and 2 years post transplant.
Incidence of Acute Graft-versus-host disease | 1 year post transplant
  Cumulative incidence of acute graft versus host disease at 1 year post transplant
Event-free survival | 1 year post transplant
  Time from transplant to death of any cause or other event, including disease relapse, graft failure, grade 3-4 acute GVHD, chronic GVHD requiring systemic therapy, or receipt of post-transplant donor cell infusion.
Disease free survival | 1 year post-transplant
  Time from transplant to death of any cause or disease relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Dimana Dimitrova, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - National Marrow Donor Program, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGAP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as the database is active.
Access Criteria: Clinical data will be made available and with permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians

REFERENCES:
- [Background] Bashey A, Zhang X, Sizemore CA, Manion K, Brown S, Holland HK, Morris LE, Solomon SR. T-cell-replete HLA-haploidentical hematopoietic transplantation for hematologic malignancies using post-transplantation cyclophosphamide results in outcomes equivalent to those of contemporaneous HLA-matched related and unrelated donor transplantation. J Clin Oncol. 2013 Apr 1;31(10):1310-6. doi: 10.1200/JCO.2012.44.3523. Epub 2013 Feb 19. PMID 23423745
- [Background] Mariotti J, Taylor J, Massey PR, Ryan K, Foley J, Buxhoeveden N, Felizardo TC, Amarnath S, Mossoba ME, Fowler DH. The pentostatin plus cyclophosphamide nonmyeloablative regimen induces durable host T cell functional deficits and prevents murine marrow allograft rejection. Biol Blood Marrow Transplant. 2011 May;17(5):620-31. doi: 10.1016/j.bbmt.2010.11.029. Epub 2010 Dec 3. PMID 21130889
- [Background] Kang E, Gennery A. Hematopoietic stem cell transplantation for primary immunodeficiencies. Hematol Oncol Clin North Am. 2014 Dec;28(6):1157-70. doi: 10.1016/j.hoc.2014.08.006. Epub 2014 Sep 16. PMID 25459185
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-C-0003.html